CLINICAL TRIAL: NCT04330833
Title: Informational Meetings for Planning and Coordinating Treatment
Acronym: IMPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Susan M Perkins, Professor of Biostatistics and Health Data Science, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1904351083; R01CA235632-01A1 (NIH)
Record Dates: First submitted 2020-02-19; First posted 2020-04-02 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-09

CONDITIONS: End of Life; Communication; Cancer Metastatic
Keywords: interventions; pediatric palliative care
MeSH Terms: conditions — Death; Communication; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: This is a multi-site, 2-group, cluster-randomized controlled trial, with clusters randomized by pediatric oncology physician-nurse dyads.
Who Masked: Participant, Outcomes Assessor
Masking Description: A trained blinded evaluator will meet with participants to complete baseline and subsequent follow-up measures, including end-of-study chart review data. Physician-nurse dyads for each arm are trained differently and naive to alternate study arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Usual Care Parent Education (Active Comparator): Parent(s) and patients receiving care from clinicians whose practice has been randomized to the enhanced usual care parent education group.
  Interventions: Other: Enhanced Usual Care Parent Education
- Novel Communication Intervention (Experimental): Parent(s) and patients receiving care from clinicians whose practice has been randomized to the novel communication intervention group.
  Interventions: Other: Novel Communication Intervention

INTERVENTIONS:
Other: Novel Communication Intervention — The intervention is a series of 3 guided discussions (using visual aids) between the child's primary oncology physician/nurse team and the child's parent(s) with the purpose of improving parental comprehension of the options for goals of treatment, along with the benefits and burdens of each option.
  Arms: Novel Communication Intervention
Other: Enhanced Usual Care Parent Education — The Enhanced Usual Care Parent Education is a series of 3 discussions between the child's primary oncology nurse and the child's parent(s) designed to control for time and attention. These discussions are focused on answering parents' questions and reviewing routine disease and treatment related information. Parents will receive a 1-hour face-to-face session every 3-4 months for a total of 3 sessions. At each session, parents choose 2-3 topics to review with the nurse.
  Arms: Enhanced Usual Care Parent Education

SUMMARY:
This prospective cluster-randomized trial examines the efficacy of a novel communication intervention delivered by trained physician and nurse dyads to parents of children with cancer within the clinicians' practice, to foster alignment of the goals of treatment. The investigators hypothesize that goal alignment will improve quality of life outcomes, in particular for those patients who reach end of life. Findings from the proposed research will provide essential information to promote communication practice standards that can be rapidly translated into practice to improve outcomes for children, particularly those who reach end of life, and parents.

DETAILED DESCRIPTION:
The overall objective of this study is to evaluate the efficacy of a novel communication intervention on quality of life outcomes in children with high-risk cancer. The intervention includes a series of tailored discussions delivered by the child's primary physician/nurse dyad that begins at diagnosis, and integrates visual aids to facilitate conversations with parents about prognosis, hopes, and goals-of-care across the cancer continuum. The central hypothesis is that the intervention will foster alignment of goals of care between providers and parents across the cancer continuum, leading to improved quality of life outcomes. Outcomes include: Enrollment in home hospice care, high-intensity medical interventions, child pain and emotional distress, parental hope, parental uncertainty and distress.

ELIGIBILITY:
Inclusion Criteria:

* Child 1 month to < 18 years
* Child newly diagnosed, i.e., within 16 weeks (112 days) from time of diagnosis of cancer not including the day of diagnosis, OR
* Child with relapsed cancer, defined as within 16 weeks (112 days) of first-time relapse/evidence of progression of disease as noted by scan or biopsy after previous diagnosis of cancer.
* Child provide assent if age ≥ 7 years
* Poor prognosis, i.e., approximate < 25 % estimated overall survival or at the discretion of the attending AND/OR:
* Falls into one of the following diagnosis categories, including but not limited to:

  * Atypical teratoid rhabdoid tumor
  * Glioblastoma multiforme
  * Diffuse intrinsic brainstem glioma
  * Embryonal tumors with multilayered rosettes
  * Other high-grade glioma
  * Gliomatosis cerebri
  * Metastatic osteosarcoma
  * Metastatic Ewing sarcoma
  * Metastatic rhabdomyosarcoma
  * Metastatic desmoplastic small round cell tumor (DSRCT)
  * Other metastatic sarcoma/carcinoma-at discretion of attending
  * Metastatic unknown primary- or rare pathology- at discretion of attending
* Parent(s) legal decision-maker(s) for child
* Parent(s) ≥18 years of age
* Parent (s) Informed of child's cancer diagnosis
* Parent(s) Able to read, speak and understand English
* Must be willing to be audio recorded during all study sessions.

Exclusion Criteria:

* The parent has neurological/cognitive impairments likely to interfere with study participation;
* The child ≥ 7 years of age does not provide assent
* Parent refuses to be audio recorded during sessions.

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 111 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Impact of Novel Communication Intervention on number of days enrolled in hospice in children with cancer and estimated 5-year survival < 25% | Within 12 months of death
  We will compare days enrolled in hospice between the Novel Communication Intervention vs Enhanced Usual Care Parent Education groups using a Wilcoxon Rank Sum Test for clustered data.

SECONDARY OUTCOMES:
Impact of the Novel Communication Intervention on the number and types of high-intensity medical interventions at end of life in children with cancer. | Within 30 days of death
  High intensity medical interventions include: code status order to attempt cardiopulmonary resuscitation, intensive care unit admission within the last 30 days, IV chemotherapy within last 14 days, greater than 2 emergency department visits within last 30 days, more than 1 hospitalization within last 30 days, not on hospice, admitted to hospice less than 3 days prior to death, intubation or cardiac resuscitation within last 30 days, and death in an acute care setting.
  The difference in the use of high-intensity medical interventions at end of life will be tested between the intervention and enhanced usual care groups with a generalized linear mixed model that accounts for subjects clustering within physician/nurse teams via a random effect.
Impact of Novel Communication Intervention on quality of life in children with cancer and estimated 5-year survival < 25% | Enrollment, then every 4 months until death or maximum of 4 years
  Quality of Life is measured with the Pediatric Quality of Life Inventory- General Module, emotional functioning sub-scale and the Pediatric Quality of Life Cancer Module. Scores range from 0-100, with higher scores indicating better health-related quality of life. Results will be modeled with linear mixed models and compared between the Novel Communication Intervention and Enhanced Usual Care Parent Education groups.
Impact of the Novel Communication Intervention on parental hope. | Enrollment, and then every 4 months until death or maximum of 4 years
  The Herth Hope Index score ranges from 12-48, with a higher score corresponding to higher levels of hope. Results from the Herth Hope Index are continuous and will be modeled with linear mixed models and compared between the intervention and enhanced usual care groups.
Impact of Novel Communication Intervention on parental adjustment to caring for a child with cancer. | Enrollment, and then every 4 months until death or maximum of 4 years
  The Parent Experience of Childhood Illness Scale (PECI)-Short Form is used to assess parental adjustment in the primary caregiver of children with chronic illness. It consists of four sub-scales with scores ranging from 0-4. Higher scores indicate poorer coping except for emotional resources, which indicates a higher level of support.
Impact of Novel Communication Intervention on parental satisfaction with healthcare | Enrollment, and then every 4 months until death or maximum of 4 years
  The Peds QL HCS (Satisfaction with Healthcare) survey is 24-item scale that measures parent satisfaction with care received from their child's oncology healthcare providers. Subscales assess parental satisfaction with:
  1. delivery of care;
  2. information received on child's diagnosis and treatments;
  3. inclusion of family;
  4. technical skills in managing their child's symptoms; and
  5. attention to their child's emotional needs.

CONTACTS AND LOCATIONS:
Overall Officials: Susan M Perkins, PhD, Principal Investigator — Indiana University
Locations (7):
- United States (7):
  - Children's Hospital Colorado, Aurora, Colorado
  - Nemours Children's Health, Wilmington, Delaware
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Riley Hospital for Children at IU Health, Indianapolis, Indiana
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - MD Anderson Children's Cancer Center, Houston, Texas
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Robb SL, Burns DS, Docherty SL, Haase JE. Ensuring treatment fidelity in a multi-site behavioral intervention study: implementing NIH Behavior Change Consortium recommendations in the SMART trial. Psychooncology. 2011 Nov;20(11):1193-201. doi: 10.1002/pon.1845. PMID 22012943
- [Background] Martin JS, Ummenhofer W, Manser T, Spirig R. Interprofessional collaboration among nurses and physicians: making a difference in patient outcome. Swiss Med Wkly. 2010 Sep 1;140:w13062. doi: 10.4414/smw.2010.13062. eCollection 2010. PMID 20458647
- [Background] Landier W, Ahern J, Barakat LP, Bhatia S, Bingen KM, Bondurant PG, Cohn SL, Dobrozsi SK, Haugen M, Herring RA, Hooke MC, Martin M, Murphy K, Newman AR, Rodgers CC, Ruccione KS, Sullivan J, Weiss M, Withycombe J, Yasui L, Hockenberry M. Patient/Family Education for Newly Diagnosed Pediatric Oncology Patients. J Pediatr Oncol Nurs. 2016 Nov/Dec;33(6):422-431. doi: 10.1177/1043454216655983. Epub 2016 Jul 9. PMID 27385664
- [Background] Horner S, Rew L, Torres R. Enhancing intervention fidelity: a means of strengthening study impact. J Spec Pediatr Nurs. 2006 Apr;11(2):80-9. doi: 10.1111/j.1744-6155.2006.00050.x. PMID 16635187
- [Background] Foster Akard T, Gerhardt CA, Hendricks-Ferguson V, Given B, Friedman DL, Hinds PS, Gilmer MJ. Facebook Advertising To Recruit Pediatric Populations. J Palliat Med. 2016 Jul;19(7):692-3. doi: 10.1089/jpm.2016.0128. Epub 2016 May 3. No abstract available. PMID 27139113
- [Background] Sawin KJ, Montgomery KE, Dupree CY, Haase JE, Phillips CR, Hendricks-Ferguson VL. Oncology Nurse Managers' Perceptions of Palliative Care and End-of-Life Communication. J Pediatr Oncol Nurs. 2019 May/Jun;36(3):178-190. doi: 10.1177/1043454219835448. Epub 2019 Apr 3. PMID 30939966
- [Background] Hendricks-Ferguson VL, Cherven BO, Burns DS, Docherty SL, Phillips-Salimi CR, Roll L, Stegenga KA, Donovan Stickler M, Haase JE. Recruitment strategies and rates of a multi-site behavioral intervention for adolescents and young adults with cancer. J Pediatr Health Care. 2013 Nov-Dec;27(6):434-42. doi: 10.1016/j.pedhc.2012.04.010. Epub 2012 Jun 2. PMID 22658379
- [Background] Hendricks-Ferguson VL, Haase JE. Parent Perspectives of Receiving Early Information About Palliative and End-of-Life Care Options From Their Child's Pediatric Providers. Cancer Nurs. 2019 Jul/Aug;42(4):E22-E30. doi: 10.1097/NCC.0000000000000589. PMID 29620556
- [Background] Hendricks-Ferguson VL, Ruebling I, Sargeant DM, Kienstra K, Eliot KA, Howell TG, Sebelski CA, Moore KS, Armstrong K. Undergraduate students' perspectives of healthcare professionals' use of shared decision-making skills. J Interprof Care. 2018 Jul;32(4):481-489. doi: 10.1080/13561820.2018.1443912. Epub 2018 Mar 7. PMID 29513119
- [Background] Hendricks-Ferguson VL, Pradhan K, Shih CS, Gauvain KM, Kane JR, Liu J, Haase JE. Pilot Evaluation of a Palliative and End-of-Life Communication Intervention for Parents of Children With a Brain Tumor. J Pediatr Oncol Nurs. 2017 May/Jun;34(3):203-213. doi: 10.1177/1043454216676836. PMID 27920233
- [Background] Hendricks-Ferguson V. Physical symptoms of children receiving pediatric hospice care at home during the last week of life. Oncol Nurs Forum. 2008 Nov;35(6):E108-15. doi: 10.1188/08.onf.e108-e115. PMID 18980914
- [Background] Hendricks-Ferguson VL, Kane JR, Pradhan KR, Shih CS, Gauvain KM, Baker JN, Haase JE. Evaluation of Physician and Nurse Dyad Training Procedures to Deliver a Palliative and End-of-Life Communication Intervention to Parents of Children with a Brain Tumor. J Pediatr Oncol Nurs. 2015 Sep-Oct;32(5):337-47. doi: 10.1177/1043454214563410. Epub 2015 Jan 26. PMID 25623029
- See also: National Cancer Institute Resource: Children with cancer: A parents' guide. — https://www.cancer.gov/publications/patient-education/guide-for-parents